CLINICAL TRIAL: NCT02882074
Title: Does Plasma Volume Replacement With 5% Human Albumin Reduce Endothelial Injury and Glycocalyceal Disruption Compared With 6% Hydroxyethylstarch (130/0.4) in Patients Having Cardiac Surgery? A Substudy of the SHARP Clinical Trial
Brief Title: Endothelial Function After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 16-342
Record Dates: First submitted 2016-08-17; First posted 2016-08-29 (Estimated); Results first posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Endothelial Dysfunction
MeSH Terms: interventions — Serum Albumin, Human; Albumins; Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Human albumin (Other): Human albumin 5% during surgery.
  Interventions: Drug: Human albumin
- Hydroxyethyl starch (Other): Hydroxyethyl starch 6% (130/0.4) solution during surgery
  Interventions: Drug: Hydroxyethyl starch

INTERVENTIONS:
Drug: Human albumin — human albumin 5% during surgery
  Other Names: albumin
  Arms: Human albumin
Drug: Hydroxyethyl starch — 6% Hydroxyethyl starch 130/0.4 during surgery
  Other Names: HES
  Arms: Hydroxyethyl starch

SUMMARY:
The purpose of this study is to evaluate whether patients receiving human albumin for plasma volume replacement during cardiac surgery have improved postoperative endothelial function compared to patients receiving 6% hydroxyethyl starch solutions. The postoperative endothelial function, measured with peripheral arterial tonometry as reactive hyperemia index (RHI) within 2 hours following surgery, will be compared in cardiac surgical patients randomized to receive human albumin or 6% HES solutions for intraoperative volume replacement. Within two hours of arrival to the ICU peripheral arterial tonometry using EndoPAT will be performed. In a subset of 40 consecutive patients the investigators will perform additional EndoPAT measurements to describe the expected changes that occur in endothelial function during the perioperative period (baseline, early postoperative and 24 hours postoperative) using RHI.

This study will also determine whether human albumin 5% reduces plasma biomarkers of endothelial and glycocalyceal damage by measuring plasma concentrations of syndecan 1 and endocan at baseline (before surgery), and 1 and 24 hours following surgery. Blood samples will be taken on the morning of the surgery, within one hour of arrival to the intensive care unit (ICU), and 24 hours after surgery or within 2 hours before discharge from the ICU (three times altogether). These samples will be used to measure the plasma concentrations of two biomarkers that measure endothelial injury.

DETAILED DESCRIPTION:
Cardiac surgical patients enrolled in the SHARP study will be randomized to 5% human albumin or 6% HES on entrance to the operating room. Anesthetic and Surgical management will follow protocol established by SHARP study including administration of a blinded study solution which contains 5% human albumin or 6% HES following separation from cardiopulmonary bypass. Blood will collected for measurement of baseline syndecan 1 and endocan following arterial line and urinary catheter placement before surgical incision. At 1 and 24 hrs following surgery completion, blood will be collected for measurement of syndecan 1 and endocan. Within two hours of ICU arrival, assessment of endothelial function will be performed.

In a subset of patients (patients who consent for multiple measurements), assessment of endothelial function will be performed preoperatively (baseline) and 24 hours after surgery.

Vasoactive substances may influence EndoPAT measurement. Thus the investigators will collect data on use of preoperative antihypertensive medications that have direct or indirect effect on arterial smooth muscle relaxation. Use of epinephrine, norepinephrine, vasopressin, milrinone, nitroglycerine, nitroprusside, and sedatives such as propofol, dexmedetomidine and others will be recorded and adjusted for in the analysis. Data on packed red blood cells (PRBC) and blood component transfusion will be collected from Anesthesia Record Keeping System. Indications for PRBC transfusion include hematocrit (HCT) <22% on cardiopulmonary bypass and <24% off cardiopulmonary bypass, and hypovolemia with anemia (HCT<25% with mean arterial blood pressure <60 mmHg or heart rate >100 bpm). Blood component transfusion (platelets, fresh frozen plasma, cryoprecipitate) may be administered as necessary following institutional standard of care. Imbalances in blood product transfusion between study groups will be adjusted for in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 - 85 years old
* Scheduled for elective aortic valve replacement with or without coronary artery bypass grafting with or without additional minor surgical procedure.
* Written, informed consent for participation in this investigation.

Exclusion Criteria:

* Patients with Raynaud's disease or other disease associated with upper extremity vascular insufficiency,
* Inability to perform EndoPAT exam (inability to lie still for 15 min, or significant finger deformity),
* Patients with renal failure with oliguria or anuria not related to hypovolemia.
* Patients receiving dialysis.
* Patients with preoperative renal insufficiency (Creatinine > 1.6 mg/dL)
* Anticipated deep hypothermic circulatory arrest
* Known hypersensitivity or allergy to hydroxyethyl starch or the excipients of hydroxyethyl starch
* Clinical conditions with volume overload (e.g., patients in pulmonary edema or congestive heart failure)
* Patients with severe hypernatremia or severe hyperchloremia
* Patients with intracranial bleeding
* Pregnant or breast feeding women
* Critically ill adult patients, including patients with sepsis, due to increased risk of mortality and renal replacement therapy, (e.g. patients who are hospitalized in the intensive care unit prior to surgery)
* Severe liver disease
* Pre-existing coagulation or bleeding disorders
* Any contraindications to proposed interventions.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2016-06; Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sessler, M.D., Study Chair — Department Chair
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Human Albumin | Hydroxyethyl Starch
Started | 43 | 42
Completed | 43 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Human Albumin | Hydroxyethyl Starch | Total
Number analyzed (Participants) | 43 | 42 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (7) | 68 (10) | 69 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 25 | 26 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 41 | 38 | 79
  Not White | 2 | 4 | 6
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 30 (5) | 30 (6) | 30 (4)

OUTCOME MEASURES:

1. Primary Outcome: Reactive Hyperemia Index (RHI)
Description: RHI measures endothelial dysfunction using noninvasive peripheral arterial tonometry (PAT) with the EndoPAT device. It is a ratio of the post-to-pre occlusion PAT amplitude of the tested arm, divided by the post-to-pre occlusion ratio of the control arm. RHI less than 1.67 is considered a sign of endothelial dysfunction and RHI equal to or greater than 1.67 is considered normal function. Increasing score indicates the improvement of coronary endothelial function.
Time Frame: 2 hours after surgery
Population: The primary endpoint, the Reactive Hyperaemia Index measured within 2 hours of ICU arrival, was missing in 12 patients from the albumin group and 8 patients from the HES group, related to the inability to obtain good quality Reactive Hyperaemia Index measurement most commonly due to movement or other artifacts. The missing primary endpoint was independent of randomization (p=0.34).
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Human Albumin | Hydroxyethyl Starch
Number analyzed (Participants) | 31 | 34
ratio | 1.88 (0.80) | 1.61 (0.71)
Statistical Analysis 1: Comparison: Human Albumin vs Hydroxyethyl Starch; Test type: Superiority; p = 0.158, Regression, Linear; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.11 to 0.64]

2. Secondary Outcome: Plasma Concentrations of Syndecan
Description: Blood samples will be obtained at specified times
Time Frame: 1 hour after surgery, 24 hours after surgery
Population: Of 141 patients in the primary clinical trial (NCT02192502), 85 patients consented to the measurement of the Reactive Hyperaemia Index. For secondary outcomes, laboratory markers were measured in the initial 141 patients (N=72 albumin, 69 hydroxyethyl starch). Syndecan 1 hour after surgery was missing in 3 patients from the albumin group and 3 patients from the HES group. Syndecan 24 hours after surgery was missing in 4 patients from the albumin group and 4 patients from the HES group.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Human Albumin | Hydroxyethyl Starch
Number analyzed (Participants) | 69 | 66
ng/mL
  Syndecan 1 hour after surgery | 684 [307 to 1249] | 746 [391 to 1499]
  Syndecan 24 hours after surgery: number analyzed (Participants) | 68 | 65
  Syndecan 24 hours after surgery | 282 [94 to 846] | 344 [102 to 1071]
Statistical Analysis 1: Comparison: Human Albumin vs Hydroxyethyl Starch; Test type: Superiority; p = 0.388, Mixed Models Analysis — The significance criterion is p-value < 0.025 (i.e. 0.05/2), corrected for multiple comparisons; Ratio of geometric means = 0.86, 97.5% CI 2-sided [0.57 to 1.28] — Syndecan values were all log-transformed to meet the linearity requirement. Thus the treatment effect was presented as the ratio of geometric means

3. Secondary Outcome: Plasma Concentrations of Endocan
Description: Blood samples will be obtained at specified times
Time Frame: 1 hour after surgery, 24 hours after surgery
Population: Of 141 patients in the primary clinical trial (NCT02192502), 85 patients consented to the measurement of the Reactive Hyperaemia Index. For secondary outcomes, laboratory markers were measured in the initial 141 patients (N=72 albumin, 69 hydroxyethyl starch). Endocan 1 hour after surgery was missing in 1 patient from the albumin group and 2 patients from the HES group. Endocan 24 hours after surgery was missing in 3 patients from the albumin group and 4 patients from the HES group.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Human Albumin | Hydroxyethyl Starch
Number analyzed (Participants) | 71 | 67
pg/mL
  endocan 1 hour after surgery | 280 [163 to 451] | 233 [158 to 444]
  endocan 24 hours after surgery: number analyzed (Participants) | 69 | 65
  endocan 24 hours after surgery | 154 [70 to 323] | 132 [51 to 333]
Statistical Analysis 1: Comparison: Human Albumin vs Hydroxyethyl Starch; Test type: Superiority; p = 0.257, Mixed Models Analysis — The significance criterion is p-value < 0.025 (i.e. 0.05/2), corrected for multiple comparisons; Ratio of geometric means = 1.19, 97.5% CI 2-sided [0.84 to 1.68] — Endocan values were all log-transformed to meet the linearity requirement. Thus the treatment effect was presented as the ratio of geometric means

4. Other Pre Specified Outcome: Reactive Hyperemia Index (RHI)
Description: as for outcome 1
Time Frame: 24 hours after surgery
Population: The secondary endpoint, the Reactive Hyperaemia Index measured within 24 hours of ICU arrival, was missing in 19 patients from the albumin group and 21 patients from the HES group, related to the inability to obtain good quality Reactive Hyperaemia Index measurement most commonly due to movement or other artifacts.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Human Albumin | Hydroxyethyl Starch
Number analyzed (Participants) | 24 | 21
ratio | 2.22 (0.68) | 1.60 (0.62)
Statistical Analysis 1: Comparison: Human Albumin vs Hydroxyethyl Starch; Test type: Superiority; p = 0.003, Regression, Linear; Mean Difference (Final Values) = 0.62, 95% CI 2-sided [0.23 to 1.01]

ADVERSE EVENTS:
Time Frame: 24 hours after surgery
Arm/Group | Human Albumin | Hydroxyethyl Starch
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/42
Other Adverse Events (participants affected / at risk) | 0/43 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT02882074/Prot_SAP_000.pdf
  • Informed Consent Form (2016-03-04): https://cdn.clinicaltrials.gov/large-docs/74/NCT02882074/ICF_001.pdf